CLINICAL TRIAL: NCT02379767
Title: Effects of Electroconvulsive Therapy on Monoamine Oxidase A Distribution Volume in Treatment-Resistant Depression Investigated With PET
Brief Title: Effects of ECT on Monoamine Oxidase A in Depression Investigated With PET
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Rupert Lanzenberger, Assoc. Prof. PD Dr. med., Medical University of Vienna
Other Study IDs: v1.2_201502
Record Dates: First submitted 2015-03-01; First posted 2015-03-05 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Major Depression
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Patients: Subjects aged between 18 and 60 years suffering from unipolar severe depression, who did not respond to conventional pharmacological antidepressant treatment (at least two adequate trials with antidepressants of different pharmacological classes over a minimum period of one month, equivalent to 150mg of tricyclic antidepressants). Concomitant psychotropic medication will be accepted during study participation, however, medication should remain stable throughout the study. Patients will undergo 6 to 14 ECT sessions in accordance with recent consensus statements and based on standard operation procedures (SOPs) of the Department of Psychiatry and Psychotherapy.
  Interventions: Device: Electroconvulsive therapy; Other: Positron emission tomography of the brain using [11C]harmine; Other: Structural magnetic resonance imaging
- Healthy subjects: Subjects will be age- and sex-matched to the patients and should present no psychiatric, or major neurological or internistic illness.
  Interventions: Other: Positron emission tomography of the brain using [11C]harmine; Other: Structural magnetic resonance imaging

INTERVENTIONS:
Device: Electroconvulsive therapy
  Groups: Patients
Other: Positron emission tomography of the brain using [11C]harmine
Other: Structural magnetic resonance imaging

SUMMARY:
This study aims at evaluating the effect of electroconvulsive therapy in treatment-resistant depressed patients on the major serotonin degrading enzyme in the human brain using neuroimaging methods, the monoamine oxidase A. Electroconvulsive therapy is an effective treatment option in severe cases of depression. However, the mechanisms underlying its effect remain uncertain, though variations within the serotonergic neurotransmitter system seem to be crucially involved.

DETAILED DESCRIPTION:
In treatment-resistant depression, electroconvulsive therapy (ECT) has been shown to effectively reduce depressive symptoms; however, the underlying neurobiological mechanisms remain to be fully understood. Recent neuroimaging findings underline the involvement of the serotonergic system in the mechanism of action of ECT, but studies in this context mainly focused on serotonin receptor and the serotonin transporter. Here, the aim of the study is to assess the effects ECT on monoamine oxidase A (MAO-A), the main serotonin degrading enzyme which is known to be involved in antidepressant action, in humans using positron emission tomography (PET) and the radiotracer [11C]harmine. Moreover, as the antidepressant effects of electroconvulsive stimulations were shown to be partly mediated via changes in neuroplasticity, a secondary aim of the present study is to assess structural alterations caused by ECT using magnetic resonance imaging (sMRI).

Based on the literature, the investigators expect higher baseline MAO-A distribution volumes (DVs) in depressed patients than compared to healthy subjects.Moreover, the investigators expect overall MAO-A distribution volume (DVs) changes in the brain of depressed patients following ECT according to the individual treatment-response. Similarly, the investigators assume that depressed patients will exhibit structural changes of grey matter volume following ECT.

The investigation is designed as a longitudinal mono-centre study over a duration of 36 months. 18 subjects with therapy-resistant, severe unipolar depression, aged between 18-60 years and 18 age- and sex-matched healthy subjects will be included in the study. Patients will be recruited at the Department of Psychiatry and Psychotherapy, Medical University of Vienna, and will be offered inpatient care. Psychotropic medication (except for drugs directly binding MAO-A, e.g. moclobemid) of the patients is allowed if steady state has been reached > 10 days prior to inclusion. Healthy subject will be recruited using announcements of poster boards at the General Hospital of Vienna. Each patient will be measured three times using a GE Advance PET scanner and the radioligand [11C]harmine. The first and second measurements determine baseline changes in the MAO-A DVs while the third scan is used to quantify changes induced by ECT. Healthy subjects will be measured with PET only once. Similarly, patients will undergo three structural (T1-weighted) MRI sessions temporally coordinated to the PET scans. Healthy subjects will be measured with MRI only once.

Each patient will be treated in 6 to 14 ECT sessions within a time interval of 2 to 5 weeks. A brief pulse ECT machine (Thymatron System IVTM) will be used three times per week to administer treatments either unilaterally over the right hemisphere or, if required, bilaterally.

The MAO-A DVs will be determined using a region of interest and a whole brain voxel-wise approach. A repeated-measures analysis of variance (ANOVA) will compare the change in the MAO-A DVs before and after ECT (PET2-PET3) with the change between the baseline PET scans (PET1-PET2). Secondly, MAO-A DVs from PET1 will be compared to the scans of healthy subjects (cross-sectional part). Additionally, the correlation between treatment effects reflected in HAM-D score and changes in MAO-A DVs will be computed. Similar statistical analyses will be done with sMRI data.

This study would be the first to demonstrate an effect of ECT on MAO-A DVs in humans in vivo. Given the involvement of the MAO-A in the pathophysiology of mood disorders, the present study would be an important step towards a better understanding of antidepressant treatment and treatment response. By comparing treatment effects and the underlying biological mechanism, the study might help to identify biomarkers that distinguish patients who are likely to benefit from ECT from patients who will rather be non-responders. Finally, by investigating the role of the MAO-A DVs in ECT, its highly discussed relevance for antidepressant action will be further elucidated and might prepare the ground for new therapeutic strategies. Additionally, this study might contribute in substantiating potential effects of ECT on brain structure.

ELIGIBILITY:
Inclusion Criteria (for patients):

* Male or female
* Age 18 - 60 years
* ICD-10 diagnosis of severe unipolar depression (ICD-10: F32.2, F32.3; F33.2, F33.3)
* A score of 23 or greater on the 17-item HAM-D
* Signed informed consent form
* Negative urine pregnancy test in women at the screening visit and at PET/MRI days
* Antidepressant and antipsychotic medication in a steady state for at least 10 days prior to inclusion
* Anesthesiological approval for ECT
* Relatively stable mental state which allows for a potential latency period of 10 days until inclusion as concomitant medication must be in steady-state for a minimum of 10 days prior ECT.

Inclusion criteria (for healthy subjects):

* Male or female
* Age 18 - 60 years
* Somatic health based on history, physical examination, ECG, and laboratory screening
* A maximum of 7 points on the 17-item HAM-D
* Signed informed consent form
* Negative urine pregnancy test in women at the screening visit and at PET/MRI days

Exclusion Criteria:

* Concomitant major internistic or neurological illness
* Clinically relevant abnormalities on a general physical examination and routine laboratory screening
* Current substance abuse, including nicotine
* Current or past history of schizophrenia or schizoaffective disorder
* For participants who participated in an earlier neuroimaging study using ionizing radiation, the total radiation exposure dose of 20 mSv over the last 10 years must not be exceeded, as specified in the legislation on radiation protection (Allg. Strahlenschutzverordnung 2010; www.ris.bka.gv.at).
* Presence of any metallic implant contraindicated for MRI
* Previous treatments with electroconvulsive therapy
* Treatment (< 1 months before screening) with bright light therapy
* Treatment (< 1 months before screening) with drugs directly affecting the density and/or activity of monoamine oxidase A, e.g. moclobemid.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 18 patients with severe unipolar depression determined by a structured clinical interview for DSM-IV (SCID) and the 17-item Hamilton Rating Scale for Depression (HAM-D score ≥ 23) who did not respond to conventional pharmacological antidepressant treatment (at least two adequate trials with antidepressants of different pharmacological classes over a minimum period of one month, equivalent to 150mg of tricyclic antidepressants) will be recruited at the Department of Psychiatry and Psychotherapy at the General Hospital of Vienna. Additionally, 18 healthy age- and sex-matched controls will participate in this longitudinal study.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2015-03; Primary Completion 2018-05-25 (Actual); Study Completion 2018-05-25 (Actual)

PRIMARY OUTCOMES:
Monoamine oxidase A distribution volume in the brain | 5 weeks
  MAOA DVs will be assessed using positron emission tomography

SECONDARY OUTCOMES:
Grey matter volume | 5 weeks
  Grey matter volume will be assessed using structural magnetic resonance imaging

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry and Psychotherapy, Vienna, Austria

REFERENCES:
- [Derived] Gryglewski G, Baldinger-Melich P, Seiger R, Godbersen GM, Michenthaler P, Klobl M, Spurny B, Kautzky A, Vanicek T, Kasper S, Frey R, Lanzenberger R. Structural changes in amygdala nuclei, hippocampal subfields and cortical thickness following electroconvulsive therapy in treatment-resistant depression: longitudinal analysis. Br J Psychiatry. 2019 Mar;214(3):159-167. doi: 10.1192/bjp.2018.224. Epub 2018 Nov 16. PMID 30442205